CLINICAL TRIAL: NCT00336687
Title: Study of Incidence, of Mechanisms and Prognosis of the Thrombopenia From Patients of Reanimation.
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Moulins Hospital (Other); Centre Hospitalier Universitaire de Saint Etienne (Other); LA ROCHE SUR YON HOSPITAL (Unknown)
Responsible Party: Fabrice Thiollière, CHU Clermont-Ferrand
Other Study IDs: CHU63-0013
Record Dates: First submitted 2006-06-13; First posted 2006-06-14 (Estimated); Last update posted 2010-03-29 (Estimated); Status verified 2010-03

CONDITIONS: Thrombopenia
Keywords: Thrombopenia; Reanimation; Thrombopenia in reanimation
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
About 40 % of the patients in reanimation are thrombopenics and the causes are not well known (reduction in platelet's production, increase in their destruction...). This protocol studies the epidemiology of thrombopenia for these patients and the impacts of cost and mortality in order to bring patients best medical cares.

DETAILED DESCRIPTION:
About 40 % of the patients in reanimation are thrombopenics and the causes are not well known (reduction in platelet's production, increase in their destruction...). This protocol studies the epidemiology of thrombopenia for these patients and the impacts of cost and mortality in order to bring patients best medical cares.

ELIGIBILITY:
Inclusion Criteria:

* Thrombopenia in reanimation

Exclusion Criteria:

* Pregnancy
* Contraindication of myelogram

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of Reanimation
Sampling Method: Non-Probability Sample
Enrollment: 322 (Estimated)
Dates: Start 2005-07; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Epidemiology of Thrombopenia and its consequences. | in reanimation

SECONDARY OUTCOMES:
The impact of cost and mortality of Thrombopenia in reanimation. | in reanimation

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Thiolliere, Dr, Study Director — University Hospital, Clermont-Ferrand
Locations (1):
- Clermont-Ferrand University Hospital, Clermont-Ferrand, Auvergne, France